CLINICAL TRIAL: NCT05029414
Title: EnDovascular Therapy Plus Best Medical Treatment (BMT) Versus BMT Alone for MedIum VeSsel Occlusion sTroke - a prAgmatic, International, Multicentre, Randomized triaL (DISTAL)
Brief Title: EnDovascular Therapy Plus Best Medical Treatment (BMT) Versus BMT Alone for MedIum VeSsel Occlusion sTroke
Acronym: DISTAL
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Basel, Switzerland (Other)
Collaborators: Swiss National Fund for Scientific Research (Other); Stryker Neurovascular (Industry); Penumbra Inc. (Industry); Medtronic (Industry); Phenox GmbH (Industry); Rapid Medical (Industry); Gottfried und Julia Bangerter- Rhyner-Stiftung, Basel (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2021-01692; qu20Psychogios2
Record Dates: First submitted 2021-08-26; First posted 2021-08-31 (Actual); Last update posted 2024-12-24 (Actual); Status verified 2024-12

CONDITIONS: Acute Ischemic Stroke
Keywords: Stroke; Medium Vessel Occlusion; Endovascular Therapy
MeSH Terms: conditions — Ischemic Stroke; Stroke

STUDY DESIGN:
Intervention Model Description: Pragmatic, parallel group, randomized, open label, superiority trial with blinded endpoint assessment
Who Masked: Outcomes Assessor
Masking Description: A treatment-blinded person will assess the primary outcome dependency and disability in everyday life (measured with the modified Rankin Scale (mRS)) at 90 days. All interviewers will be certified for the conductance of mRS.
  interviews.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group: EVT + BMT (Experimental): Patients randomized to the EVT arm will undergo endovascular therapy (EVT) in addition to best medical treatment (BMT). All decisions regarding EVT device and EVT technique will be made by the treating physician.
  Interventions: Procedure: Endovascular Therapy
- Control group: BMT (No Intervention): Patients randomized to the control arm will NOT undergo EVT but will get best medical treatment (BMT) including intravenous thrombolysis (IVT) or antiplatelet therapy if indicated under current international guidelines and according to routine clinical practice.

INTERVENTIONS:
Procedure: Endovascular Therapy — Endovascular treatment of stroke is the non-surgical treatment for the sudden loss of brain function due to blood clots. The blood clot is removed from the blood via devices (i.e. stent-retriever, aspiration catheters and balloon guide) to achieve revascularization.
  Arms: Intervention group: EVT + BMT

SUMMARY:
Acute ischemic stroke (AIS) is one of the main causes of disability and loss of quality adjusted life years. This study is to analyze whether endovascular therapy (EVT) in addition to best medical treatment (BMT) reduces the degree of disability and dependency in daily activities after a Medium Vessel Occlusion (MeVO) stroke compared to BMT alone.

DETAILED DESCRIPTION:
Acute ischemic stroke (AIS) is one of the main causes of death and disability and thereby the third leading cause of loss of quality adjusted life years. For patients with an AIS due to an occlusion of the large vessels of the anterior circulation, endovascular therapy (EVT) has become a treatment standard. 20-40% of all AIS patients have occlusions of smaller vessels and present with a more distal isolated Medium Vessel Occlusion (MeVO). The primary objective of this randomized trial is to determine whether patients experiencing an AIS due to an isolated medium vessel occlusion have superior functional outcome (measured with the Modified Rankin Scale "mRS" at 90 days) when treated with EVT plus best medical treatment (BMT) compared to patients treated with BMT alone. In this trial, all commercially available, CE-certified revascularisation devices (i.e. stent-retriever, aspiration catheters and balloon guide catheters) can be used for EVT. All established techniques for the endovascular treatment of AIS patients are permitted and all decisions regarding treatment technique and choice of devices and/or medications are made solely by the treating physician.

ELIGIBILITY:
Inclusion Criteria:

* Acute ischemic stroke
* Treatment (arterial puncture) can be initiated 2.1. Within 6 hours of last seen well (LSW) OR 2.2. Within 6 to 24 hours of LSW AND
* CT Criteria: Evidence of a hypoperfusion-hypodensity mismatch (Absence of hypodensity on the noncontrast CT within ≥ 90% of the area of the hypoperfused lesion on perfusion CT)
* MRI Criteria: Evidence of a diffusion-hyperintensity mismatch (Absence of hyperintensity on fluid-attenuated inversion recovery (FLAIR) imaging within ≥ 90% of the area of the diffusion weighted imaging(DWI) lesion)
* Isolated medium vessel occlusion (i.e. an occlusion of the co-/non-dominant M2, the M3/M4 segment of theMCA, the A1/A2/A3 segment of the ACA or the P1/P2/P3 segment of the PCA) confirmed by CT or MRIAngiography
* National Institute of Health Stroke Scale (NIHSS) Score of ≥ 4 points or symptoms deemed clearly disabling by treating physician (i.e. aphasia, hemianopia, etc.)
* Informed Consent as documented by signature or fulfilling the criteria for emergency consent/ deferral consent
* Agreement of treating physician to perform endovascular procedure

Exclusion Criteria:

* Acute intracranial haemorrhage
* Patient bedridden or presenting from a nursing home
* In-Hospital Stroke
* Known (serious) sensitivity to radiographic contrast agents, nickel, titanium metals or their alloys
* Foreseeable difficulties in follow-up due to geographic reasons (e.g. patients living abroad)
* Pregnancy or lactating women. A negative pregnancy test before randomisation is required for all women with child-bearing potential.
* Known history of arterial tortuosity, pre-existing stent, other arterial disease and/or known disease at the arterial access site that would prevent the device from reaching the target vessel and/or preclude safe recovery after EVT
* Severe comorbidities, which will likely prevent improvement or follow-up
* Radiological confirmed evidence of mass effect or intracranial tumour (except small meningioma)
* Radiological confirmed evidence of cerebral vasculitis
* Evidence of vessel recanalization prior to randomisation
* Participation in another interventional trial

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 543 (Actual)
Dates: Start 2021-12-09 (Actual); Primary Completion 2024-10-10 (Actual); Study Completion 2025-06-01 (Estimated)

PRIMARY OUTCOMES:
Degree of dependency and disability in everyday life (measured with the mRS) | at 90 days (± 14 days) after randomisation
  The primary outcome is the degree of dependency and disability in everyday life (measured with the mRS) at 90 days. The mRS is the standard tool to assess neurological outcome in trials with acute severe brain disease. The scale runs from 0-6, running from perfect health without symptoms (= 0) to death (= 6).

SECONDARY OUTCOMES:
Change in National Institutes of Health Stroke Scale (NIHSS) | 24 hours post-randomization (+/- 6 hours)
  The scale is made up of 11 different elements that evaluate specific ability. The score for each ability is a number between 0 and 4, 0 being normal functioning and 4 being completely impaired. The patient's NIHSS score is calculated by adding the number for each element of the scale; 42 is the highest score possible. In the NIHSS, the higher the score, the more impaired a stroke patient is.
Assessment of Cognitive function using the validated Montreal cognitive assessment (MoCA) | at 90 days (± 14 days) after randomisation
  MoCA scores range between 0 and 30. A score of 26 or over is considered to be normal.
Change in Quality of life as assessed by the EuroQol-5D | at 90 ± 14 days and at 1 year after randomisation
  The EQ-5D descriptive system comprises five dimensions: mobility, self-care, usual activities, pain and discomfort, and anxiety and depression.
  the descriptive system produces a 5-digit health status profile that represents that person's level of reported problems on the five EQ-5D health dimensions
Degree of dependency and disability in everyday life (measured with the mRS) | at one year (± 30 days) after randomisation
  Degree of dependency and disability in everyday life (measured with the mRS). The scale runs from 0-6, running from perfect health without symptoms (= 0) to death (= 6).
Patient residential status | at one year (± 30 days) after randomisation
  Patient residential status will be obtained through a telephone call to the patient or if not available his next of kin/caregiver one year (± 30 days) after randomisation
Change in percentage of penumbral tissue saved (Imaging Data Evaluation) | at baseline and post-interventional at 24 hours (± 6 hours) post-randomisation
  Percentage of penumbral tissue saved (Imaging Data Evaluation): It is defined as the proportion of tissue at risk (defined as the mismatch volume derived from with RAPID Compute tomography perfusion (CTP) (IschemaView Inc.) at baseline that did not progress to infarction at 24h (derived from Magnet Resonance Imaging (MRI) (FLAIR and Diffusion Weighted Imaging (DWI)) or NCCT imaging.
Radiologic occurrence of intracranial haemorrhages | within 24 hours (± 6 hours) post randomisation
  Radiologic occurrence of intracranial haemorrhages graded according to the modified Safe Implementation of Thrombolysis in Stroke-Monitoring Study (SITS-MOST) definition

OTHER OUTCOMES:
Change in All-cause mortality (Safety Outcome) | at days 7-10 or discharge if earlier, 90 day ± 14 days; and one year ± 30 days after randomisation.
  Change in All-cause mortality
Change in Serious Adverse Events (SAEs) | at 24 h ± 6h, days 7-10 or discharge if earlier and at 90 ± 14 days after randomisation
  Change in Serious Adverse Events (SAEs)
Change in symptomatic intracranial haemorrhage | at 24 ± 6 hours post randomisation
  Change in symptomatic intracranial haemorrhage by radiologic categorization on the basis of the pre-randomisation imaging at day 0 (Non contrast computed tomography (NCCT)/Magnet Resonance Imaging (MRI), Computed tomography angiography (CTA)/Magnetic Resonance Angiography (MRA), Diffusion Weighted Imaging (DWI)/Perfusion Weighted Imaging (PWI) MRI, Compute tomography (CT) perfusion) and the post-interventional imaging at 24 ± 6 hours.

CONTACTS AND LOCATIONS:
Overall Officials: Marios-Nikos Psychogios, Prof.Dr., Principal Investigator — Department of Interventional and Diagnostical Neuroradiology, University Hospital Basel; Urs Fischer, Prof.Dr., Principal Investigator — Neurology, Inselspital, Bern University Hospital
Locations (56):
- Belgium (6):
  - AZ Sint-Jan Brugge, Bruges
  - Hôpital Civil Marie Curie Charleroi, Charleroi
  - UZ Universiteit Gent, Ghent
  - AZ Groeninge, Kortrijk
  - Universitair Ziekenhuis Leuven, Leuven
  - Clinique CHC MontLégia, Liège
- Finland (2):
  - Helsinki University Hospital, Helsinki
  - Turku University Hospital, Turku
- Germany (15):
  - Uniklinik RHTW Aachen, Aachen
  - Charité-Universitätsmedizin Berlin, Berlin
  - Klinikum Bremen-Mitte, Bremen
  - Uniklinikum Dresden, Dresden
  - Helios Klinikum Erfurt, Erfurt
  - University Hospital Frankfurt, Frankfurt
  - University Medical Center Göttingen, Göttingen
  - Asklepios Klinik Altona, Hamburg, Hamburg
  - University Hospital Hamburg Eppendorf, Hamburg
  - University Medical Center Mannheim, Mannheim
  - Universitätsklinikum der Technischen Universität München, München
  - University Hospital Münster, Münster
  - Klinikum Nürnberg, Nuremberg
  - Klinikum VEST GmbH, Recklinghausen
  - Klinikum der Landeshauptstadt Stuttgart gKAöR, Stuttgart
- Hadassah-Hebrew University Medical Center, Jerusalem, Israel
- Italy (4):
  - Maggiore Hospital, Bologna
  - Careggi University Hospital,, Florence
  - Antonio Cardarelli Hospital, Napoli
  - San Giovanni Bosco Hospital, Torino
- Netherlands (8):
  - Amsterdam University Medical Center, Amsterdam
  - Rijnstate Hospital Arnhem, Arnhem
  - University Medical Center Groningen, Groningen
  - Leiden University Medical Center, Leiden
  - Maastricht University Medical Center, Maastricht
  - Radboud University Medical Center Nijmegen, Nijmegen
  - Erasmus MC University Medical Center Rotterdam, Rotterdam
  - Haaglanden Medical Center, The Hague
- Lisbon Central University Hospital, Lisbon, Portugal
- Spain (7):
  - Hospital Clinico Barcelona, Barcelona
  - Hospital Vall d'Hebron, Barcelona
  - University Hospital Germans Trias i Pujol, Barcelona
  - University Hospital Doctor Josep Trueta, Girona, Girona
  - University Hospital Clínico San Carlos, Madrid, Madrid
  - University Hospital Virgen de la Arrixaca, Murcia, Murcia
  - Hospital Clinico Universitario de Valladolid, Valladolid
- Skane University Hospital, Lund, Sweden
- Switzerland (10):
  - Kantonsspital Aarau, Department of Interventional and Diagnostical Neuroradiology, Aarau
  - Department of Interventional and Diagnostical Neuroradiology, Clinic of Radiology and Nuclear Medicine, University Hospital Basel, Basel
  - Department of Neurology, University Hospital Basel, Basel
  - Inselspital Bern, University Clinic for Neuroradiology, Bern
  - Geneva University Hospitals, Interventional Neuroradiology Unit, Geneva
  - Centre hospitalier universitaire vaudois, CHUV, Lausanne
  - Kantonsspital Luzern, Lucerne
  - Neurocentro (EOC) della Svizzera Italiana Stroke Center, Servizio di Neurologia, Ospedale Civico, Lugano
  - Kantonsspital St Gallen, Sankt Gallen
  - University Hospital Zurich, Departement of Neuroradiology, Zurich
- Barts NHS Health Trust, London, United Kingdom

REFERENCES:
- [Background] Marios-Nikos P, Alex B, Jens F, Isabel F, Jan G, Mira K, Ronen L, Paolo M, Marc R, Jeffrey L S, Daniel S, Adriaan VE, Claus Z, Nikki R, Luzia B, Urs F. EnDovascular therapy plus best medical treatment (BMT) versus BMT alone for medIum distal veSsel occlusion sTroke (DISTAL): An international, multicentre, randomized-controlled, two-arm, assessor-blinded trial. Eur Stroke J. 2024 Dec;9(4):1083-1092. doi: 10.1177/23969873241250212. Epub 2024 May 3. PMID 38702876
- [Derived] Psychogios M, Brehm A, Ribo M, Rizzo F, Strbian D, Raty S, Arenillas JF, Martinez-Galdamez M, Hajdu SD, Michel P, Gralla J, Piechowiak EI, Kaiser DPO, Puetz V, Van den Bergh F, De Raedt S, Bellante F, Dusart A, Hellstern V, Khanafer A, Parrilla G, Morales A, Kirschke JS, Wunderlich S, Fiehler J, Thomalla G, Lemmens R, Peluso JP, Bolognese M, von Hessling A, van Es A, Kruyt ND, Coutinho JM, Castano C, Minnerup J, van Zwam W, Dhondt E, Nolte CH, Machi P, Loehr C, Mattle HP, Buhk JH, Kaesmacher J, Dobrocky T, Papanagiotou P, Alonso A, Holtmannspoetter M, Zini A, Renieri L, Keil F, van den Wijngaard I, Kagi G, Terceno M, Wiesmann M, Amaro S, Rommers N, Balmer L, Fragata I, Katan M, Leker RR, Saver JL, Staals J, Fischer U; DISTAL Investigators. Endovascular Treatment for Stroke Due to Occlusion of Medium or Distal Vessels. N Engl J Med. 2025 Apr 10;392(14):1374-1384. doi: 10.1056/NEJMoa2408954. Epub 2025 Feb 5. PMID 39908430